CLINICAL TRIAL: NCT04738318
Title: Steroid Administration for Articular Fractures of the Elbow (SAFE Trial): A Randomized, Controlled Trial of Perioperative Glucocorticoids During Treatment of Intraarticular Elbow Fractures
Brief Title: Steroid Administration for Articular Fractures of the Elbow (SAFE Trial)
Acronym: SAFE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Switched to observational study type.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jed Maslow, Assistant Professor, Department of Orthopaedic Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210125
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Elbow Fracture
Keywords: Glucocorticoid Administration
MeSH Terms: conditions — Elbow Fractures | interventions — Glucocorticoids; Dexamethasone; Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treating physician and patient will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Glucocorticoid) (Experimental): Patients will receive a single intraoperative dose of 10mg of intravenous dexamethasone. Following surgery, the participant will be provided with a 1) six-day oral methylprednisolone taper course.
  Interventions: Drug: Glucocorticoids
- Control Arm (Placebo) (Placebo Comparator): Patients will receive a single intraoperative dose of 10 mg of saline. Following surgery, the participant will be provided with a six-day placebo course.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Glucocorticoids — Patients will receive a single intraoperative dose of 10mg of intravenous dexamethasone intraoperatively. Following surgery, the participant will be provided with a six-day oral methylprednisolone taper course.
  Other Names: Dexamethasone; Methylprednisolone
  Arms: Treatment Arm (Glucocorticoid)
Drug: Saline — Patients will receive a single intraoperative dose of 10 mg of saline. Following surgery, the participant will be provided with a six-day placebo course.
  Arms: Control Arm (Placebo)

SUMMARY:
The primary purpose of this study is to determine if perioperative glucocorticoid administration (IV intra-operative followed by a post-operative oral taper course) improves post-operative range of motion in a patient population that has sustained an intra-articular elbow fracture(s) (radial head, proximal ulna, distal humerus, or combined) that required operative fixation.

DETAILED DESCRIPTION:
Elbow fractures are complex injuries that often involve the articular surface, are in close proximity to critical neurovascular structures, and are prone to post-operative complications. Complications following treatment of intra-articular elbow pathology can affect over 50% of patients and up to 30% of all patients will require a re-operation. One of the most common complications is joint stiffness.1 When a flexion arc of motion is diminished to less than 100 degrees, a flexion contracture is present greater than 30 degrees, or forearm rotation is less than 100 degrees, functional limitations are frequently present and further treatment may be recommended.2,3 In fact, contracture release may be required in 12-20% of patients after intra-articular elbow fractures and carries a relatively high complication rate when performed.

The relationship of post-traumatic elbow contracture to intra-articular fractures is well established and can caused by extrinsic factors such as heterotopic ossification (HO), fibrosis and capsular thickening, or by intrinsic factors such as failure of nonunion, malunion, arthrosis, or loose bodies.2,4 Recent studies analyzing the acute phase synovial fluid cytokine profile after an intra-articular elbow fracture have shown proinflammatory and catabolic factors in high concentrations that can lead to contracture through myofibroblast differentiation and proliferation.4 Furthermore, HO can limit range of motion in up to 40% of fractures and may also result from prolonged inflammation with elevated IL-1β and TNF-α levels.

The purpose of this study is to determine if perioperative glucocorticoid administration (IV intra-operative followed by a post-operative oral taper course) improves post-operative range of motion in a patient population that has sustained an intra-articular elbow fracture(s) (radial head, proximal ulna, distal humerus, or combined) that required operative fixation.

Primary Study Questions

1. For adult patients (>18yo) who sustain intra-articular elbow fractures (radial head, proximal ulna, distal humerus, or combined) that undergo operative fixation, does perioperative glucocorticoid administration (IV intra-operative followed by a post-operative oral taper course) improve post-operative range of motion (flexion/extension and pronation/supination) compared to a placebo?

   Secondary Study Questions
2. Is perioperative glucocorticoid administration more effective in improving range of motion for certain intra-operative elbow fractures or depending on the mechanism of injury (subgroup comparison based on fracture type and high-energy or low-energy injuries)?
3. Do patients that receive perioperative glucocorticoids have a higher surgical site infection rate?

ELIGIBILITY:
Inclusion Criteria

• All adults ≥18 years old with an isolated, intra-articular traumatic elbow fracture to be treated at Vanderbilt University Medical Center with operative intervention and a standardized post-operative rehab protocol.

* Intra-articular elbow fracture defined as:

  * Distal humerus
  * Proximal ulna
  * Radial head fracture
  * Combination fracture of two or more of the above
* Radiographs present confirming intra-articular injury

Exclusion Criteria

* Patients with bilateral elbow fractures
* Patients with an altered mental status
* Pregnant
* Allergy or contra-indication to glucocorticoid administration
* Type 1 or Type 2 diabetes
* Pre-injury limitation in elbow range or motion (patient reported)
* Unable to provide consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Chen HW, Liu GD, Wu LJ. Complications of treating terrible triad injury of the elbow: a systematic review. PLoS One. 2014 May 15;9(5):e97476. doi: 10.1371/journal.pone.0097476. eCollection 2014. PMID 24832627
- [Background] Kodde IF, van Rijn J, van den Bekerom MP, Eygendaal D. Surgical treatment of post-traumatic elbow stiffness: a systematic review. J Shoulder Elbow Surg. 2013 Apr;22(4):574-80. doi: 10.1016/j.jse.2012.11.010. Epub 2013 Feb 1. PMID 23375881
- [Background] Morrey BF, Askew LJ, Chao EY. A biomechanical study of normal functional elbow motion. J Bone Joint Surg Am. 1981 Jul;63(6):872-7. PMID 7240327
- [Background] Wahl EP, Lampley AJ, Chen A, Adams SB, Nettles DL, Richard MJ. Inflammatory cytokines and matrix metalloproteinases in the synovial fluid after intra-articular elbow fracture. J Shoulder Elbow Surg. 2020 Apr;29(4):736-742. doi: 10.1016/j.jse.2019.09.024. Epub 2019 Nov 26. PMID 31784384
- [Background] Desai MJ, Matson AP, Ruch DS, Leversedge FJ, Aldridge JM 3rd, Richard MJ. Perioperative Glucocorticoid Administration Improves Elbow Motion in Terrible Triad Injuries. J Hand Surg Am. 2017 Jan;42(1):41-46. doi: 10.1016/j.jhsa.2016.11.011. PMID 28052827
- [Background] Kaneguchi A, Ozawa J, Yamaoka K. Anti-inflammatory Drug Dexamethasone Treatment During the Remobilization Period Improves Range of Motion in a Rat Knee Model of Joint Contracture. Inflammation. 2018 Aug;41(4):1409-1423. doi: 10.1007/s10753-018-0788-5. PMID 29911276
- [Background] Wu Y, Lu X, Ma Y, Zeng Y, Bao X, Xiong H, Shen B. Perioperative multiple low-dose Dexamethasones improves postoperative clinical outcomes after Total knee arthroplasty. BMC Musculoskelet Disord. 2018 Dec 1;19(1):428. doi: 10.1186/s12891-018-2359-1. PMID 30501618
- [Background] Xu H, Zhang S, Xie J, Lei Y, Cao G, Pei F. Multiple Doses of Perioperative Dexamethasone Further Improve Clinical Outcomes After Total Knee Arthroplasty: A Prospective, Randomized, Controlled Study. J Arthroplasty. 2018 Nov;33(11):3448-3454. doi: 10.1016/j.arth.2018.06.031. Epub 2018 Jul 4. PMID 30033064
- [Background] Pugh DM, Wild LM, Schemitsch EH, King GJ, McKee MD. Standard surgical protocol to treat elbow dislocations with radial head and coronoid fractures. J Bone Joint Surg Am. 2004 Jun;86(6):1122-30. doi: 10.2106/00004623-200406000-00002. PMID 15173283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One of the enrolled participants was withdrawn following consent but prior to study randomization because their treating physician decided post-consent the participant required a different surgery which made the participant ineligible to participate in the study.
Period: Overall Study
Arm/Group | Treatment Arm (Glucocorticoid) | Control Arm (Placebo)
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were no participants randomized to the control arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm (Glucocorticoid) | Control Arm (Placebo) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 30 [23 to 37] |  | 30 [23 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m2] | 25.6 [23.8 to 27.5] |  | 25.6 [23.8 to 27.5]

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Range of Motion of Elbow
Description: Flexion, extension, pronation, supination
Time Frame: Change between 2-week, 6-week, 3-month, 6-month, and final follow-up visits.
Population: Data analysis was not completed because only one participant completed the Treatment arm and zero patients completed the Control arm. Disclosing the data could violate privacy interests.
Arm/Group | Treatment Arm (Glucocorticoid) | Control Arm (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Serious Adverse Event- Any untoward medical occurrence that results in death or is life-threatening, results in persistent or substantial disability or incapacitation, results in inpatient hospitalization, or prolongation of an existing hospitalization, or requires medical or surgical intervention to prevent any of the previously mentioned outcomes as a result of this research.
  Adverse Event Collection- An adverse event log was completed at each post-operative timepoint by study personnel.
Arm/Group | Treatment Arm (Glucocorticoid) | Control Arm (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early and converted to a non-interventional, observational study model. Of the 3 participants consented prior to termination, only 2 were randomized to a treatment arm and only 1 completed study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT04738318/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT04738318/SAP_001.pdf